CLINICAL TRIAL: NCT04982172
Title: Model-informed Infliximab Dose De-escalation Following Earlier Dose Escalation in Adult Patients With Inflammatory Bowel Diseases
Brief Title: Model-informed Dose De-escalation of Infliximab in Patients With Inflammatory Bowel Diseases
Acronym: MODIFI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S64521
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2022-02

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Infliximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional arm (Experimental): Model-informed precision dosing of infliximab (intravenously administered) using a Bayesian forecasting software tool. Doses and dosing intervals will be derived from the software tool, aiming to maintain adequate exposure (trough concentration target 5 mg/L).
  Interventions: Drug: Infliximab
- Historical control arm (Active Comparator): The treating physician adjusted the intravenously administered infliximab doses and dosing intervals without being guided by a model-informed precision dosing software tool. The primary objective was to extend the dosing interval. Therefore, dose de-escalation (interval extension with/without dose adjustment) were performed following a scheme at the treating physician's discretion.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Infliximab (Inflectra® [Pfizer]), dosage determined using model-informed precision dosing, intravenously administered
  Arms: Interventional arm
Drug: Infliximab — Infliximab, dosage following a dose de-escalation algorithm at the physician's discretion, intravenously administered
  Arms: Historical control arm

SUMMARY:
This is a monocentric, two-arm, non-randomised, non-blinded, historically controlled, interventional trial. The purpose of this trial is to investigate the effect of model-informed infliximab dose de-escalation on the infliximab exposure and therapeutic outcome as compared to standard dose de-escalation in patients with inflammatory bowel diseases.

ELIGIBILITY:
Inclusion Criteria:

* The subject or, when applicable, the subject's legally acceptable representative signs and dates a written informed consent form and any required privacy authorisation prior to the initiation of any study procedures.
* The subject is aged 18 to 80 years inclusive.
* The subject has a good understanding of the Dutch language.
* The subject is diagnosed with moderately to severely active ulcerative colitis or Crohn's disease, confirmed by clinical, endoscopic, histological, and/or imaging criteria.
* The subject was in maintenance therapy, later lost their response to treatment and subsequently gained steroid-free, clinical and biological remission following infliximab dose escalation (i.e., by increasing the dose and/or shortening the dosing interval) and had an infliximab trough concentration ≥5 mg/L.
* Adequate contraception in female subjects of reproductive age (oral contraception, intra-uterine device, sterilisation or barrier method).

Exclusion Criteria:

* The subject is aged <18 years or >80 years.
* The subject receives infliximab prophylactically (e.g. in the immediate postoperative setting).
* The subject has an ostomy or an ileal anal pouch anastomosis.
* If female subjects, when pregnant (based on a positive serum sample) or lactating or intending to become pregnant or nurse before, during or within 15 weeks after the last dose of study drug; or intending to donate ova during such time period.
* The subject is participating in another interventional clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Steroid-free, combined clinical and biological remission | During one year after start of infliximab dose de-escalation
  The proportion of patients maintaining steroid-free, combined clinical and biological remission during one year after infliximab dose de-escalation based on a standard dosing algorithm versus a model-informed dosing algorithm.
  Combined clinical and biological remission is defined based on patient-reported outcomes (rectal bleeding score = 0 + stool frequency score ≤1 [ulcerative colitis], mean daily abdominal pain score ≤1 + liquid stool frequency score ≤1.5 [Crohn's disease]) together with normal C-reactive protein (<5 mg/L) and faecal calprotectin (<250 mg/kg). Steroid-free indicates the absence of any dose of any oral or rectal steroid use.

SECONDARY OUTCOMES:
Steroid-free, combined clinical and biological remission | At one year after start of infliximab dose de-escalation
  The proportion of patients maintaining steroid-free, combined clinical and biological remission at one year after infliximab dose de-escalation based on a standard dosing algorithm versus a model-informed dosing algorithm.
  Combined clinical and biological remission is defined based on patient-reported outcomes (rectal bleeding score = 0 + stool frequency score ≤1 [ulcerative colitis], mean daily abdominal pain score ≤1 + liquid stool frequency score ≤1.5 [Crohn's disease]) together with normal C-reactive protein (<5 mg/L) and faecal calprotectin (<250 mg/kg). Steroid-free indicates the absence of any dose of any oral or rectal steroid use.

OTHER OUTCOMES:
Steroid-free clinical remission | At and during one year after start of infliximab dose de-escalation
  The proportion of patients maintaining steroid-free clinical remission at and during one year after infliximab dose de-escalation based on a standard dosing algorithm versus a model-informed dosing algorithm.
  Clinical remission is defined based on patient-reported outcomes (rectal bleeding score = 0 + stool frequency score ≤1 [ulcerative colitis], mean daily abdominal pain score ≤1 + liquid stool frequency score ≤1.5 [Crohn's disease]).
  Steroid-free indicates the absence of any dose of any oral or rectal steroid use.
Steroid-free biological remission | At and during one year after start of infliximab dose de-escalation
  The proportion of patients maintaining steroid-free biological remission at and during one year after infliximab dose de-escalation based on a standard dosing algorithm versus a model-informed dosing algorithm.
  Biological remission is defined as normal C-reactive protein (<5 mg/L) and faecal calprotectin (<250 mg/kg).
  Steroid-free indicates the absence of any dose of any oral or rectal steroid use.
Infliximab trough concentration target attainment and area under the concentration-time curve | At and during one year after start of infliximab dose de-escalation
  Exposure: Trough concentration (target attainment; 5 mg/L) and area under the concentration-time curve.
Total infliximab dose and number of infusions | At and during one year after start of infliximab dose de-escalation
  Dosage: total infliximab dose (# mg) and number of infusions.
Direct costs calculated based on cost of infliximab and cost related to the day hospital needed for the infusion | At one year after start of infliximab dose de-escalation
  Direct costs calculated based on cost of infliximab and cost related to the day hospital needed for the infusion (in euro).
Indirect costs based on questionnaire | At one year after start of infliximab dose de-escalation
  Indirect costs based on questionnaire: iMTA Productivity Cost Questionnaire (iMTA PCQ)
Health-related quality of life based on QoL questionnaire | At one year after start of infliximab dose de-escalation
  Health-related quality of life based on QoL questionnaire: Inflammatory Bowel Disease Questionnaire (IBDQ-32)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ferrante, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Flanders, Belgium

REFERENCES:
- [Derived] Kantasiripitak W, Outtier A, Wicha SG, Kensert A, Wang Z, Sabino J, Vermeire S, Thomas D, Ferrante M, Dreesen E. Multi-model averaging improves the performance of model-guided infliximab dosing in patients with inflammatory bowel diseases. CPT Pharmacometrics Syst Pharmacol. 2022 Aug;11(8):1045-1059. doi: 10.1002/psp4.12813. Epub 2022 Jun 15. PMID 35706358